CLINICAL TRIAL: NCT06036628
Title: National Surveillance of the Use of New Antibiotics in Pediatrics and Multi- Resistant Bacteria Involved in Pediatric Infections
Brief Title: Resistant Bacteria in Children in France
Acronym: BREF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: BREF
Record Dates: First submitted 2023-04-28; First posted 2023-09-14 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-09

CONDITIONS: Infection Due to Resistant Bacteria; Multi-antibiotic Resistance; Antibiotic Prescription; Risk Factors; Healing; Complications; Intensive Care Unit; Hospital Discharge; Outcome, Fatal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is observational, multicenter and prospective study for surveillance of the use of new antibiotics in pediatrics for treated pediatrics infections due to multi-resistant bacteria

DETAILED DESCRIPTION:
The main of this study is to evaluate the relevance of prescribing "new antibiotics" according to the antibiogram of the isolated bacteria or in the absence of bacteriological documentation

As this is a surveillance study, the clinical and biological characteristics of the children included will be described.

ELIGIBILITY:
Inclusion Criteria:

* Children under 18 years of age
* Hospitalized in France in a hospital center working with the ACTIV/GPIP network
* Treated with one or more of the following antibiotics:

  * Colimycin (Colistimethate sodium)
  * Cefiderocol
  * Aztreonam in combination
  * Ceftolozane-Tazobactam
  * Ceftazidime-avibactam
  * Meropenem/vaborbactam
  * Imipenem/Relebactam
  * Tigecycline
  * Daptomycin
  * Ceftaroline fosamil
  * Tedizolid phosphate
  * Fidaxomicin
  * Ceftobiprole
  * Dalbavancin

In association with a documented infection performed by:

* Blood culture
* Normally sterile site

  * Cerebrospinal fluid
  * Pleural fluid
  * Pleura
  * Peritoneum
  * Joint fluid
  * Other
* Urine sampling if the bacteria was considered responsible for the infection (associated with a leukocyturia ≥10,0000)
* Respiratory specimens if the bacteria was considered responsible for the infection
* Sampling on material such as:Intubation probe, Orthopedic, Urological, Central Nervous System (CNS),....

  * Related to colonization with multidrug-resistant bacteria without documentation.

Exclusion Criteria:

* Refusal of participation by the patient or his/her parent
* Medical history of mucoviscidosis

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatrics patients infected by multi-resistant bacterial, treated by new antibiotics
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Relevance of prescribing "new antibiotics" according to patient status | 1 year
  Type of new antibiotics prescribed for pediatrics infections caused by multi-resistant bacteria according to the antibiogram of the isolated bacteria or in the absence of bacteriological documentation
Relevance of prescribing "new antibiotics" | 1 year
  how are used new antibiotics prescribed for pediatrics infections caused by multi-resistant bacteria

SECONDARY OUTCOMES:
Describe Bacterial epidemiology of infections associated with prescription of new antibiotics | 1 year
  Characteristic of bacteria associated with prescription of new antibiotics
Identify Risks factors for multi-resistant bacteria | 1 year
  Type of conditions responsible of multi-resistant such as comorbidities, travel, previous hospitalization, previous antibiotherapy,
Describe Context of drug Prescription | 1 year
  How antibiotics medical prescriptions are controlled and validated
Department involved in medical prescribing | 1 year
  Number of department involved in medical prescriptions
Describe Associated Antibiotherapies type | 1 year
  Type of drug association prescribed
Describe Associated Antibiotherapies | 1 year
  Number of drug association prescribed
Describe patients outcome | 1 year
  Proportion of patients clinically and bacteriologically recovered

CONTACTS AND LOCATIONS:
Overall Officials: Levy Corinne, Study Director — Association Clinique Thérapeutique Infantile du val de Marne; Cohen Robert, Principal Investigator — Association Clinique Thérapeutique Infantile du val de Marne
Locations (1):
- ACTIV, Créteil, France